CLINICAL TRIAL: NCT06971601
Title: Diagnostic Validity of Infrapatellar Fat Pad Impingement Syndrome: Performance of Clinical Tests Compared to MRI Imaging
Brief Title: Diagnostic Validity Ofclinical Tests for Infrapatellar Fat Pad Impingement Syndrome
Acronym: ETICHOFFA
Status: Not yet recruiting | Type: Observational
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Other Study IDs: ETICHOFFA; 2024-A02410-47 (Other: ANSM)
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Anterior Knee Pain
Keywords: Hoffa's fat pad; Infrapatellar fat pad; Diagnosis; MRI
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Provocative test — The clinical evaluation specific to Infrapatellar fat pad is based on a series of five standardized clinical tests, extensively described in the specialized literature: provoked palpation of the fat pad, provoked passive extension, Hoffa's test, gliding test, and provoked passive flexion. These tests are performed in a randomized order to limit sequence bias. A test is considered positive if it reproduces the patient's typical anterior knee pain with an intensity greater than 2/10 on the numerical pain scale. Although widely used, these tests have not yet undergone rigorous methodological validation, which this study specifically aims to address.

SUMMARY:
The ETICHOFFA study is a clinical research project aiming to improve the diagnosis of Infrapatellar fat pad impingement syndrome, a common source of anterior knee pain. Although MRI remains the gold standard for diagnosis, clinical testing strategies lack validation. This observational study has two main objectives: to assess the diagnostic accuracy of a cluster of standardized clinical provocation tests for IFP impingement compared to MRI findings, and to identify clinical and subjective characteristics associated with IFP involvement confirmed by imaging.

This observational study will recruit 50 patients aged 18 to 70 years with anterior knee pain rated at least 3 out of 10 in intensity. Participants will complete a secure online questionnaire documenting symptoms, pain distribution, aggravating and relieving factors, and pain intensity at rest, during activity, and daily life. They will also complete three validated scales: the Anterior Knee Pain Scale (AKPS), the Knee injury and Osteoarthritis Outcome Score (KOOS), and the Tampa Scale for Kinesiophobia (TSK).

A standardized clinical examination will be performed, including subpatellar skin temperature measurement, knee swelling assessment, passive range of motion testing, and a series of provocation tests targeting Hoffa's fat pad. Tests will be randomized to reduce bias and considered positive if they reproduce the patient's typical pain with an intensity of at least 2/10. Each participant must also undergo a standardized MRI of the knee within two weeks of the clinical assessment, interpreted blindly by an independent musculoskeletal radiologist.

All data will be anonymized, stored securely, and analyzed using SPSS software. Diagnostic accuracy of clinical tests will be evaluated through sensitivity, specificity, predictive values, and likelihood ratios. Functional outcomes related to taping will also be analyzed.

The study has received ethical approval and adheres to GDPR standards for data protection. Participation is voluntary, with the right to withdraw at any time. The ETICHOFFA study is expected to enhance clinical diagnostic pathways for anterior knee pain associated with Infrapatellar fat pad involvement.

DETAILED DESCRIPTION:
Study Protocol Description The ETICHOFFA study is a clinical research project aiming to improve the diagnosis of infrapatellar fat pad (IFP) impingement syndrome, a common but under-recognized source of anterior knee pain. Although magnetic resonance imaging (MRI) remains the diagnostic gold standard, clinical testing strategies for IFP involvement are poorly standardized and lack validated diagnostic performance.

This observational study has two main objectives: (1) to assess the diagnostic accuracy of a cluster of standardized clinical provocation tests for IFP impingement compared to MRI findings, and (2) to identify clinical and subjective characteristics associated with IFP involvement confirmed by imaging.

The sample size of 50 participants was determined by an a priori power calculation. The primary hypothesis is that a composite score based on five clinical provocation tests will yield an area under the ROC curve (AUC) of at least 0.80, a threshold commonly considered indicative of good diagnostic discrimination. The null hypothesis is set at an AUC of 0.50, representing no discriminative ability. Using a two-sided alpha level of 0.05 and a statistical power of 80% (1-β), and assuming a prevalence of positive MRI findings of approximately 33% (i.e., a 2:1 ratio of test negatives to positives), the number of positive cases required was estimated at 11, corresponding to a total of 33 participants (11 positives and 22 negatives). Accounting for a 10% anticipated loss or exclusion rate, the total sample size was increased to 37 participants. However, this calculation is based on idealized assumptions and does not fully capture the uncertainties inherent to clinical research under real-world conditions. Variability in actual IFP prevalence, incomplete or uninterpretable MRI data, and interindividual variability in clinical test responses may all affect the study's effective statistical power. Therefore, a sample size of 50 participants was ultimately planned to ensure robust analysis and compensate for such contingencies.

The study will proceed in the following steps:

Step 1: Patient Inclusion Patients will be eligible if they are aged between 18 and 70 years and experience anterior knee pain with an intensity of ≥ 3/10 on a numerical pain scale on most days over the past month.

Certain medical conditions will be exclusion criteria, including: recent corticosteroid injections (within 12 months), hip or back surgery, specific neurological conditions, and any contraindications to MRI.

Prior to enrollment, each patient will receive detailed information and have the opportunity to ask any questions. Informed written consent will be obtained.

Step 2: Clinical Evaluation Each participant will complete a secured online questionnaire (GDPR-compliant platform) to record symptoms, painful areas (via bodychart), aggravating and relieving factors, and pain intensity (via visual analogue scale [VAS]/100) at rest, during physical activity, and in everyday situations. Three validated functional questionnaires (AKPS, KOOS-PF and Tampa scale Kinesiophobia) will also be completed to assess the impact of pain on daily activities and quality of life.

The clinical examination will be performed by a team of three physiotherapists and three physical medicine and rehabilitation (PM&R) physicians, all trained across two standardized theoretical sessions. These sessions will cover both the study procedures and the standardized execution and interpretation of the clinical tests. All examiners will be blinded to the MRI results and to participants' self-reported data in order to minimize assessment bias. A standardized clinical examination will be conducted, including measurement of infrapatellar skin temperature using an infrared thermometer, assessment of knee swelling via the stroke test, passive knee range of motion (flexion and extension), and a set of five clinical tests targeting IFP. These include provocative palpation, passive extension and flexion tests, Hoffa's test, and IFP gliding test (a mobility assessment scored on a three-level ordinal scale: hypomobile, normal, or hypermobile). All tests will be performed in randomized order to minimize examiner bias and will be considered positive if they reproduce the patient's typical pain with an intensity of at least 2/10.

Step 3: Knee MRI A knee MRI must have been performed within two weeks before or after the clinical evaluation.

The MRI will follow a standardized protocol including T1 and T2 sequences, allowing the detection of Hoffa's fat pad abnormalities (inflammation, fibrosis, hypertrophy).

Interpretations will be carried out by an independent radiologist blinded to the clinical findings to ensure objective assessment.

Step 4: Data Processing and Analysis The clinical test results will be compared to MRI findings. Following data collection, a random sample of 33 participants will be selected a posteriori for the primary diagnostic accuracy analysis. This post hoc randomization is intended to reduce selection bias, overfitting, and spectrum bias, by ensuring that the analysis is not influenced by knowledge of the final diagnostic outcome or distribution of positive and negative cases. Diagnostic performance (both individual and combined tests) will be evaluated through: Sensitivity, Specificity, Predictive values, Likelihood ratios, Overall discriminative ability and post-test probability estimates using Fagan nomograms.Recognized statistical methods (notably SPSS software) will be used, and all analyses will be conducted blinded to group assignments.

All collected information will remain strictly confidential and anonymized. Data will be coded using a unique identifier (e.g., the first three letters of the last name plus date of birth) and stored in a secured Excel file accessible only to the research team.

The study's total duration is estimated at 12 months, with a 6-month inclusion period. Participation involves a single session, during a regular consultation with a physiotherapist or physician. No particular restrictions will apply regarding participation in other studies in parallel.

The ETICHOFFA study is expected to improve the clinical diagnostic pathway for anterior knee pain by validating simple clinical tests to detect infrapatellar fat pad impingement in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Presence of anterior knee pain with an intensity of ≥3/10 on the Numerical Rating Scale (NRS), on most days over the past month
* MRI of the knee performed within a maximum of 15 days before or after the clinical examination.

Exclusion Criteria:

* History of corticosteroid injection treatment within the previous 12 months;
* Known allergy or skin intolerance to medical adhesives or rigid tape;
* History of hip or lumbar spine surgery;
* History of neurological disorders or a diagnosis of fibromyalgia;
* Contraindication to MRI (e.g., metallic foreign body, incompatible implantable device)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 70 years experiencing anterior knee pain (AKP) rated ≥3/10 for at least 4 weeks will be eligible. Patients will be recruited from the department of orthopedic and trauma at Hôpital Paris-Est Val de Marne (Saint-Maurice), including both postoperative cases (e.g., post-arthroscopy) and non-surgical patients referred for expert consultation regarding persistent or unexplained anterior knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the diagnostic value of the five clinical tests targeting the infrapatellar fat pad, considered collectively as a test cluster. | At baseline (post-imaging and clinical assessment)
  The overall performance of the test cluster will be analyzed using contingency matrices comparing the combined clinical test results with MRI findings. Various combination strategies will be tested (e.g., ≥2 positive tests out of 5), and the following diagnostic validity indices will be calculated for each threshold: sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and positive and negative likelihood ratios (LR⁺, LR-). ROC curves will be generated, and the area under the curve (AUC) will be used as a synthetic indicator of the cluster's discriminative capacity, with an AUC ≥ 0.80 considered clinically meaningful.

SECONDARY OUTCOMES:
Diagnostic performance of individual clinical tests | At baseline (post clinical assessment)
  A set of five standardized clinical tests targeting Hoffa's fat pad will be performed on the symptomatic knee and analyzed individually against MRI findings. Four tests are pain provocation tests, and one is a mobility assessment. Diagnostic accuracy will be evaluated using sensitivity, specificity, predictive values (PPV, NPV), and likelihood ratios (LR⁺, LR-), with 95% confidence intervals. For the mobility test, ordinal logistic regression and diagnostic performance across categories will be explored.
  All tests will be conducted during the initial clinical examination. The diagnostic value of each test will be compared independently to MRI-confirmed Infrapatellar pad impingement. Unit of Measure: diagnostic accuracy metrics (Se, Sp, PPV, NPV, LR⁺, LR-); ordinal score (gliding test)
Post-test probability of Infrapatellar fat pad impingement (Fagan nomogram analysis) | At baseline (post-imaging and clinical assessment)
  To estimate the clinical decision-making utility of each provocation test, the post-test probability of Hoffa's fat pad impingement will be calculated based on positive and negative likelihood ratios (LR⁺ and LR-) derived from diagnostic performance data. A pre-test probability will be defined using the observed prevalence in the study cohort. Post-test probabilities will be determined using Bayesian reasoning and represented graphically using Fagan nomograms. This analysis aims to illustrate how individual test results impact diagnostic certainty and assist in clinical reasoning.Unit of Measure: Post-test probability (%)
Infrapatellar skin temperature at rest (lying position) | At baseline (during initial clinical assessment)
  A localized skin temperature measurement will be performed using a non-contact infrared laser thermometer, approximately 1 cm below the inferior pole of the patella (infrapatellar region). This will be the first measurement taken on the knee, about 10 minutes after the start of the consultation, with the patient in a seated position at rest. It will be performed before any physical contact with the knee, to avoid influencing local temperature.Unit of Measure: degrees celsius (°C)
Presence of intra-articular swelling (Stroke Test) | At baseline (during initial clinical assessment)
  The presence of intra-articular effusion will be assessed using the standardized Stroke Test (also known as the bulge test). The patient will be in a supine position with the knee in full extension. The examiner will use a sweeping motion to displace fluid medially and laterally around the patella. The result will be graded on a 4-point scale (0 = no wave, 1 = small wave on medial side, 2 = larger bulge, 3 = spontaneous return without sweeping). This test will be performed early in the clinical examination, before any active or passive knee mobilization.Unit of Measure: Grading scale (0 to 3)
Passive range of motion of the knee (flexion and extension) | At baseline (during initial clinical assessment)
  Passive knee flexion and extension will be assessed with the patient in a supine position, using a standard goniometer. Measurements will be taken after initial non-contact assessments (e.g., temperature and swelling evaluation) to avoid influencing resting joint status. The examiner will guide the limb through its available passive range without patient effort. The maximum flexion and extension angles (in degrees) will be recorded separately for each knee. Unit of Measure: Degrees (°)
Body Mass Index (BMI) | At baseline (during initial clinical assessment)
  BMI will be calculated using the standard formula: weight (in kilograms) divided by height (in meters) squared kg/m^2. Weight and height will be measured during the initial clinical assessment using a calibrated medical scale and stadiometer, with the patient in light clothing and without shoes.Unit of Measure: kg/m^2
Location of anterior knee pain (pain localization map) | At baseline (during initial clinical assessment)
  Patients will be asked to identify the area(s) where they experience anterior knee pain by selecting one or more standardized images depicting different anatomical zones around the patella (labelled A to F). Each image corresponds to a specific location (e.g., infrapatellar, retropatellar, medial or lateral peripatellar). Patients may select multiple images if the pain is present in more than one area. This assessment will be conducted during the clinical interview, prior to any physical examination or palpation. The responses will be categorized based on the image codes (A-I) for subsequent analysis.Unit of Measure:Categorical anatomical zones (A to I)
Anterior Knee Pain Scale (AKPS) | At baseline (during initial clinical assessment)
  The Anterior Knee Pain Scale (AKPS), also known as the Kujala score, will be used to assess perceived functional limitations related to patellofemoral disorders. The questionnaire consists of 13 items covering activities such as walking, running, squatting, and stair climbing. Scores range from 0 to 100, with higher scores indicating better knee function.
Knee Injury and Osteoarthritis Outcome Score - Patellofemoral subscale (KOOS-PF) | At baseline (during initial clinical assessment)
  The KOOS-PF subscale will be used to evaluate symptoms and functional limitations specific to patellofemoral pain. The subscale includes 11 items scored on a 5-point Likert scale. Scores are normalized from 0 to 100, with higher scores indicating fewer symptoms and better function.
Tampa Scale for Kinesiophobia (TSK-11) | At baseline (during initial clinical assessment)
  The 11-item Tampa Scale for Kinesiophobia (TSK-11) will be used to assess fear of movement or reinjury in individuals with knee pain. Each item is scored on a 4-point Likert scale, and total scores range from 11 to 44, with higher scores indicating greater fear-avoidance beliefs.
Pain intensity at rest (VAS/100) | At baseline (during initial clinical assessment)
  Pain intensity at rest will be assessed using a 100-mm visual analogue scale (VAS), where 0 represents "no pain" and 100 represents "worst imaginable pain." The measurement will be taken with the patient seated, at the beginning of the clinical evaluation.
Pain intensity during physical activity (VAS/100) | At baseline (during initial clinical assessment)
  Pain intensity during physical activity will be measured using a 100-mm visual analogue scale (VAS) immediately after patients perform standardized functional tasks (e.g., walking, stair stepping). The scale ranges from 0 ("no pain") to 100 ("worst imaginable pain").
Pain intensity in everyday situations (VAS/100) | At baseline (during clinical interview)
  Patients will rate their average pain intensity experienced in daily life over the past week using a 100-mm visual analogue scale (VAS), from 0 ("no pain") to 100 ("worst imaginable pain"). This score reflects the overall perceived burden of knee pain in everyday activities.